CLINICAL TRIAL: NCT06935773
Title: The Effectiveness of High-Fidelity Simulation-Based Emergency Scenario Training on Emergency and Critical Care Nurses' Resuscitation Knowledge and Team Resource Management Skills
Brief Title: High-Fidelity Simulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pei Yu Huang (Other)
Responsible Party: Sponsor-Investigator, Pei Yu Huang, Research Nurse Practitioner, Chang Bing Show Chwan Memorial Hospital
Organization: Chang Bing Show Chwan Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ChangBingSCMH
Record Dates: First submitted 2025-04-06; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: High-fidelity Simulation
MeSH Terms: interventions — Observation

STUDY DESIGN:
Intervention Model Description: This study adopts a quasi-experimental design, targeting the nursing staff in the emergency department and intensive care unit of Chang Bing Show Chwan Memorial Hospital for the high-fidelity simulated emergency scenario in-service training as the experimental group. The control group consists of nursing staff from the emergency and critical care units at Changhua Show Chwan Memorial Hospital. The study is conducted using a pre-test and post-test design for both groups. The measurement tools include the Team Resource Management (TRM) scale and the Emergency Knowledge scale, which are used to evaluate the training effectiveness. The experimental group is divided into subgroups based on their unit attributes and receives 20 minutes of cognitive education followed by 40 minutes of simulation training. The content includes rotating through emergency roles and post-training discussions to promote learning reflection and behavior improvement.
Who Masked: Participant
Masking Description: This study adopts a quasi-experimental design, targeting the nursing staff in the emergency department and intensive care unit of Chang Bing Show Chwan Memorial Hospital for the high-fidelity simulated emergency scenario in-service training as the experimental group. The control group consists of nursing staff from the emergency and critical care units at Changhua Show Chwan Memorial Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental - Chang Bing Show Chwan Memorial Hospital (Experimental): Participants in this group will receive high-fidelity simulated emergency scenario in-service training.
  Interventions: Other: High-Fidelity Simulated Emergency Training
- Placebo Comparator - Show Chwan Memorial Hospital (Placebo Comparator): Participants in this group will not receive any simulation-based training during the study period.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: High-Fidelity Simulated Emergency Training — A high-fidelity simulation-based in-service training program focusing on emergency scenarios. The training includes simulated resuscitation cases, teamwork drills, and post-simulation debriefings conducted at Chang Bing Show Chwan Memorial Hospital.
  Arms: Experimental - Chang Bing Show Chwan Memorial Hospital
Other: No intervention (observational study) — Participants in this arm will not receive any training or simulation intervention during the study period.
  Arms: Placebo Comparator - Show Chwan Memorial Hospital

SUMMARY:
This study explores the impact of high-fidelity simulation-based training on critical care nurses' emergency knowledge, skills, and teamwork in emergency and intensive care units. Using a quasi-experimental design, the experimental group undergoes 20 minutes of cognitive education followed by 40 minutes of simulation training, while the control group receives standard training. The study aims to assess improvements in teamwork efficiency, clinical decision-making, and confidence, with expected outcomes including enhanced emergency response skills and patient safety. The findings will underscore the value of simulation training in improving nursing care quality in high-pressure clinical environments.

DETAILED DESCRIPTION:
Research Background: Emergency departments and intensive care units (ICUs) have a high incidence of emergency events, with nurses often being the first responders to cardiac arrest situations. Therefore, they must be equipped with proficient cardiopulmonary resuscitation (CPR) skills and the ability to work effectively in emergency teams to improve survival rates.

Research Objective: This study aims to explore the impact of high-fidelity simulation-based training on enhancing the first aid skills and teamwork efficiency of critical care nurses. Additionally, it seeks to evaluate the effects of this training on nurses' emergency knowledge, skills, and ability to collaborate in emergency situations.

Research Methods: This study adopts a quasi-experimental design, targeting the nursing staff in the emergency department and intensive care unit of Chang Bing Show Chwan Memorial Hospital for the high-fidelity simulated emergency scenario in-service training as the experimental group. The control group consists of nursing staff from the emergency and critical care units at Changhua Show Chwan Memorial Hospital. The study is conducted using a pre-test and post-test design for both groups. The measurement tools include the Team Resource Management (TRM) scale and the Emergency Knowledge scale, which are used to evaluate the training effectiveness. The experimental group is divided into subgroups based on their unit attributes and receives 20 minutes of cognitive education followed by 40 minutes of simulation training. The content includes rotating through emergency roles and post-training discussions to promote learning reflection and behavior improvement.

Expected Results: It is anticipated that the high-fidelity simulation training will significantly enhance the emergency knowledge, skills, teamwork capabilities, confidence, and clinical decision-making abilities of critical care nurses.

Clinical Practice Implications: High-fidelity simulation training offers nurses the opportunity to practice in a safe environment, allowing repeated learning experiences. This approach effectively strengthens emergency response skills and teamwork, ultimately leading to improved clinical nursing quality and patient safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 years old.
2. At least three months of work experience in acute and critical care units.
3. Have received Advanced Cardiac Life Support(ACLS) training courses in hospitals.
4. Willing participants after explaining the purpose of the study.

Exclusion Criteria:

1. Nurses who are newly hired within 3 months.
2. Have not received ACLS training courses in hospitals.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
teamwork capabilities | High-fidelity simulated first aid scenarios were measured pre-intervention and post-intervention in on-the-job training
  This study used a self-developed "First Aid Knowledge Scale" based on the American Heart Association (2020) First Aid Training Guidelines and course content to evaluate the effectiveness of on-the-job training in high-fidelity simulated first aid scenarios. The scale covers core topics, including first aid and CPR concepts, medication selection and dosage, and oxygen supply frequency. To ensure content validity, five emergency specialists reviewed the scale. It consists of 10 multiple-choice questions, each with four options. Correct answers earn 1 point, and incorrect answers earn 0. The score range is 0-10, with higher scores indicating better first aid knowledge.
  The "Team Resource Management Scale" (Chen Zhijie, 2011) was used to assess teamwork before and after the intervention. It measures leadership, communication, situational monitoring, and mutual support, with a total of 33 items. Higher scores reflect better teamwork.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Bing Show Chwan Memorial Hospital, Changhua, Lukang, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
In this study, participants were divided into two groups: the experimental group (Changbin Xiuchuan) and the control group (Changhua Xiuchuan), using intentional sampling. Participants were enrolled based on specific inclusion and exclusion criteria. The experimental group was subjected to a structured intervention, while the control group did not receive the same intervention.
  The intervention for the experimental group consisted of a comprehensive on-the-job training program that simulated first aid situations. This program was designed to improve both cognitive understanding and practical skills in emergency care. Prior to the intervention, participants in the experimental group completed a pre-intervention questionnaire to assess their baseline knowledge and skills in first aid and team resource management (TRM). One week after completing the intervention, participants in the experimental group were asked to complete a post-intervention questionnaire to measure any changes in thei
Supporting Information: Study Protocol
Time Frame: one year